CLINICAL TRIAL: NCT06538272
Title: An Early Phase II, Multicenter, Placebo-Controlled, Randomized, Double-Blind, Parallel-Group, Comparison Study to Investigate the Chemotherapy-Induced Peripheral Neuropathy (CIPN) Onset-Suppressing Effect and Safety of ONO-2910 in Patients With Breast Cancer Receiving Weekly Paclitaxel
Brief Title: Study to Investigate the Chemotherapy-Induced Peripheral Neuropathy (CIPN) Onset-Suppressing Effect and Safety of ONO-2910 in Patients With Breast Cancer Receiving Weekly Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ONO-2910-03
Record Dates: First submitted 2024-07-24; First posted 2024-08-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-2910 (Experimental)
  Interventions: Drug: ONO-2910
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2910 — ONO-2910 Tablet will be orally administered once daily.
  Arms: ONO-2910
Drug: Placebo — Placebo Tablet will be orally administered once daily.
  Arms: Placebo

SUMMARY:
To investigate the safety and CIPN onset-suppressing effect of ONO-2910 in participants receiving paclitaxel (PTX) weekly as chemotherapy for breast cancer in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ECOG Performance Status 0 or 1
2. Patients scheduled to receive 12 consecutive weekly doses of PTX (80 mg/m2, intravenous infusion) as a perioperative treatment of clinical stage I-III breast cancer (concomitant use of trastuzumab and pertuzumab is allowed)
3. Patients who meet the following organ functions according to the laboratory test results at the time of treatment registration.However, blood transfusions and measurements within 7 days after administration of granulocyte colony-stimulating factor (G-CSF) are excluded.

Neutrophil count >= 1,500/mm3, Platelet count >= 75,000/mm3, Hemoglobin >= 10.0 g/dL or >= 6.2 mmol/L, Serum creatinine <= 2.0 mg/dL, Total bilirubin <= 3.0 mg/dL, ALT and AST <= 100 IU/L or less than 2.5 times the facility's upper limit of clinical laboratory test values

Exclusion Criteria:

1. Patients with grade 1 or higher peripheral sensory neuropathy, peripheral motor neuropathy, or extremity edema in the upper or lower extremities.
2. Patients with pain or numbness in the upper or lower extremities due to a history/complication, such as stroke, diabetic neuropathy, alcoholic neuropathy, carpal tunnel syndrome, tarsal tunnel syndrome, chronic inflammatory demyelinating polyradiculoneuropathy, Guillain-Barre syndrome, Fisher syndrome, knee osteoarthritis, hernia, cervical spondylosis, lumbar spondylosis, spinal canal stenosis, peripheral circulatory disorders, hand-foot syndrome,etc.
3. Patients who have difficulty in evaluating limb symptoms due to trauma/defects in the upper or lower limbs, or complications such as infectious or inflammatory diseases on the skin of the upper or lower limbs.
4. Patients with concurrent multiple cancers.
5. Patients who have not recovered from toxicity (Grade 1 or less) from prior treatment.
6. Patients who have been administered platinum agents, bortezomib, vinca alkaloids, and taxanes including PTX in the past, and patients who are scheduled to be administered these drugs other than PTX during the study period.
7. Prior treatment other than trastuzumab or pertuzumab (chemotherapy, molecular targeted drug therapy, antibody therapy, hormone therapy, immunotherapy, radiation therapy, etc.) within 7 days before the start of the treatment period (Visit 2) (including the start date of the treatment period) ) was performed.
8. At the beginning of the treatment phase (Visit 2), Patients using peripheral neuropathic pain medications such as pregabalin, mirogabalin, duloxetine, tricyclic and tetracyclic antidepressants, gabapentin, analgesics such as loxoprofen and acetaminophen, vitamin B12 such as mecobalamin, chinese herbal medicines indicated for pain such as goshajinkigan, and opioids such as oxycodone.
9. Patients who plan to receive preventive compression therapy (surgical gloves, elastic stockings, etc.) or preventive cooling therapy for chemotherapy-induced limb adverse events during the study period
10. Patients scheduled for surgery during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation：Proportion of participants with peripheral sensory neuropathy (NP)# of Grade 2 or higher by 12 weeks after the start of intervention | 12 week
Number of Participants with AE | Up to 101 days
Weight | Up to 87 days
body temperature | Up to 87 days
pulse rate | Up to 87 days
blood pressure | Up to 87 days
ECG heart rate | Up to 87 days
ECG RR interval | Up to 87 days
ECG PR interval | Up to 87 days
ECG QRS complex | Up to 87 days
ECG QT interval | Up to 87 days
ECG QTcF | Up to 87 days
Hematology | Up to 87 days
Clinical chemistry | Up to 87 days
Blood coagulation | Up to 87 days
Urinalysis | Up to 87 days
Pregnancy test | Up to 101 days
Viral test | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (30):
- Japan (30):
  - Fujita Health University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Nagoya University Hospital, Aichi
  - Funabashi Municipal Medical Center, Chiba
  - Medical Corporation Tesshokai Kameda Medical Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - Kitakyushu City Hospital Organization Kitakyushu Municipal Medical Center, Fukuoka
  - Gunma Prefectural Cancer Center, Gunma
  - University of Tsukuba Hospital, Ibaraki
  - Social Medical Corporation Hakuaikai Sagara Hospital, Kagoshima
  - Nippon Medical School Musashikosugi Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kumamoto University Hospital, Kumamoto
  - Okayama University Hospital, Okayama
  - Nahanishi Clinic, Okinawa
  - Osaka Breast Clinic, Osaka
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka
  - Osaka Rosai Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Yodogawa Christian Hospital, Osaka
  - Japanese Saitama Red Cross Hospital, Saitama
  - Saitama Medical University International Medical Center, Saitama
  - Shizuoka General Hospital, Shizuoka
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Tokyo
  - Toranomon Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No